CLINICAL TRIAL: NCT05858281
Title: Lived Experiences of Black Girls in Richmond
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM20025559
Record Dates: First submitted 2023-05-04; First posted 2023-05-15 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Lived Experiences, Strengths, and Community Assets of Black Girls
MeSH Terms: interventions — Surveys and Questionnaires; Interviews as Topic; Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Online Survey
  Interventions: Behavioral: Survey
- Focus group
  Interventions: Behavioral: Focus group
- Interviews
  Interventions: Behavioral: Interviews

INTERVENTIONS:
Behavioral: Survey — Black adolescent girls (aged 12-17) will participate in an online survey and will be asked questions regarding their strengths, family, school and community experiences, sexual education knowledge, physical health and mental wellbeing, etc.
  Groups: Online Survey
Behavioral: Interviews — Parents/guardians of Black girls (aged 12-17) and Black emerging adult women aged 18-22 will participate in individual interviews and will be asked questions about their understanding of Black girls' strengths and resources.
  Groups: Interviews
Behavioral: Focus group — Black adolescent girls (aged 12-17) will participate in a focus group and will be asked questions regarding their strengths, family, school and community resources, etc.
  Groups: Focus group

SUMMARY:
This study is to understand the quality of life of Black Girls in Richmond, Virginia, which includes generating a report about the status of Black girls in Richmond. Research or reports about the state of the girls are growing more common across the country in cities like Los Angeles, Chicago, and Philadelphia. Most of these studies generate deficit narratives focusing on these groups' problems, needs, and deficiencies. Fewer studies focus solely on the experience of Black girls specifically. This study proposes a new approach and explores the quality of life of Black girls using an asset-based approach that thinks differently about the subject of these studies and how to address their needs appropriately.

ELIGIBILITY:
Inclusion Criteria (Online Survey and focus groups):

* Self-identify as Black/African American adolescent cisgender girls, between the ages of 12-17, and reside in the City of Richmond.

Exclusion Criteria (Online Survey and focus groups):

* Girls who are not between 12 to 17 years of age, do not self-identify as Black, does not identify as cisgender, legal residence is not located in the city of Richmond, and/or who do not read English.

Inclusion Criteria (Interviews):

* Parents/guardians (any sex; no age range for parent/guardian) of Black girls (ages 12-17) who reside in the City of Richmond; and
* Black emerging adult women (ages 18-22) who resided in the City of Richmond when they were under 18.

Exclusion Criteria (Interviews):

* Parent/Guardian - Does not have a child (daughter) between the ages of 12-17; child does not self-identify as cisgender and Black/African American; legal residence is not in the city of Richmond; unable to read, write, or speak in English.
* Emerging adult women - does not self-identify as Black/African American, under 18 or over the age of 22, did not reside in the City of Richmond under 18, and unable to read, write, or speak in English.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Black girls who participate in the focus groups and online survey must self-identify as a cisgender female; and Black emerging women who participate in the interviews must self-identity as cisgender female. Parents/guardians of Black girls who participate in the interviews can be of any gender.
Study Population: Black girls aged 12-17 who self identity as cisgender girls and who live in Richmond, VA; Black emerging adult women aged 18-22 who self identify as cisgender female and who lived in Richmond, VA when they were under 18; Parents/guardians of Black girls aged 12-17 who live in Richmond, VA
Sampling Method: Non-Probability Sample
Enrollment: 339 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Survey Outcome | 3 months
  Exploration Subscale is a 7-item instrument about individuals' exploration of their ethnicity measured on a 4-point scale. Community Experience Subscale is measured by a 5-item Rasch-validated measure of youth interpersonal resilience measured on a 4-point scale. Gendered Racial Pride & Empowerment Subscale is a 19-item scale that reflect the intersectional racial and gender messages young African American women receive measured on a 4-point scale. Spiritual Support Subscale is a 13-item scale that measures spiritual maturity in persons of diverse religious and spiritual beliefs measured on a 6-point scale. Safety and Perceived Safety is a 7-item scale that measures community safety perceived measured on a 5-point scale. Physical Health & Mental Wellbeing is measured by 13 items of the 36-Item Short Form Survey measured on a 6-point scale or a 5-point scale. Sleep scale is a 5-item measure of subjective sleep quality for adolescents aged 12-18 years measured on a 6-point scale.
Focus group outcome | 3 months
  Strengths of Black girls: summarize the themes of strengths of Black girls; Community assets: summarize the themes of community assets for Black girls
Interviews outcome | 3 months
  Strengths of Black girls: summarize the themes of strengths of Black girls; Community assets: summarize the themes of community assets for Black girls

CONTACTS AND LOCATIONS:
Overall Officials: Nakeina Douglas-Glenn, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No